CLINICAL TRIAL: NCT05538208
Title: Efficacy & Safety of Pharmacokinetically-Driven Dosing of Mycophenolate Mofetil for the Treatment of Pediatric Proliferative Lupus Nephritis- A Double-Blind Placebo Controlled Clinical Trial
Brief Title: The Pediatric Lupus Nephritis Mycophenolate Mofetil (PLUMM) Study
Acronym: PLUMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Genentech, Inc. (Industry); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Hermine Brunner, MD, Division Director Rheumatology, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ML42264; 1R01AR079124-01A1 (NIH)
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-02

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Eligible patients enrolled in the study will be randomized (1:1) at baseline to the 53-week double-blind, active comparator 2-part study to receive either MMFPK or MMFBSA. Subjects who are partial renal responders (PRR) to MMFBSA at week 26, will cross over to the MMFPK arm. Complete renal responders (CRR) at week 26 in MMFBSA arm will continue to be treated with MMFBSA. Subjects with at least a PRR (or even CRR) in the MMFPK arm at week 26 will remain in the MMFPK arm and continue to receive MMF dosage targeting MPA-AUC0-12 > 60-70 mg*h/l. Subjects whose LN fails to respond to therapy by week 26 will be discontinued from the study interventions to receive LN treatment as per their local physician's decision. Subjects who experience a single episode of a LN flare during Part 1 of the study or fulfill other criteria for discontinuation from the study intervention, will also receive LN treatment as per their local physician's decision.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During this double-blinded study, the Sponsor, subject, and investigator site staff will all be blinded to the subject's treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MMFBSA (Active Comparator): MMF dosed as per body-surface area
  Interventions: Drug: Mycophenolate Mofetil
- MMFPK (Experimental): MMF dosed as per pharmacokinetically-guided precision-dosing
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — MMF dosed 600mg/m2 body surface area per dose about every 12 hours
  Other Names: MMF dosed per body surface area
  Arms: MMFBSA
Drug: Mycophenolate Mofetil — MMF dosed twice daily to achieve an area under the concentration-time curve (AUC 0-12h) of MPA >=60-70 mg*h/L
  Other Names: MMF dosed phrmacokinetically
  Arms: MMFPK

SUMMARY:
The study is a 1-year 2-part double-blinded placebo controlled 2-arm clinical trial. Treatment arms are (1) MMF dosed as per body-surface area (MMFBSA; 600mg/m2 body surface area per dose about every 12 hours) and (2) pharmacokinetically-guided precision-dosing of MMF (MMFPK; MMF dosed twice daily to achieve an area under the concentration-time curve (AUC0-12h) of MPA >60-70 mg*h/L. The study goal is to determine the safety and efficacy of MMFPK compared to MMFBSA for the treatment of proliferative LN in subjects 8 to <21 years.

DETAILED DESCRIPTION:
Subjects will be randomized 1:1 to receive blinded treatment with MMFPK or MMFBSA for up to 53 weeks. The primary endpoint, clinical remission of LN, is measured at the end of Part 1 at week 26. Subjects in the MMFBSA arm who have only partial renal response (PRR) at the end of Part 1 will newly receive MMFPK upon entering Part 2 of the study (week 26 - 53). Subjects with complete renal responses (CRR) at the end of Part 1 will continue the same dosing regimen of MMF (MMFBSA or MMFPK) in Part 2 as was given in Part 1 of the study. Subjects in the MMFPK arm with PRR at the end of Part 1 will enter Part 2 and continue in the MMFPK arm.

Subjects who are LN non-responders by the end of Part 1 at week 26 will be considered treatment failures and discontinued from the study intervention. All subjects who are discontinued from the study intervention for reasons of efficacy or safety will receive LN treatment and monitoring as per the treating physician's decision. However, these subjects will be asked to participate in study visits at weeks 26 and 53/End of Study.

ELIGIBILITY:
Inclusion

1. Male or female aged 8 to < 21 years;
2. Must meet Classification Criteria for SLE as per the criteria of the American College of Rheumatology (ACR)/ European League Against Rheumatism
3. Diagnosed with proliferative LN as per the International Society of Nephrology/Renal Pathology Society4 based on kidney biopsy done within 90 days prior to enrollment into the study;

   Subjects may have been previously diagnosed with LN. For study inclusion, the kidney biopsy must be interpreted as one of the following classes: Class 3, Class 3/5, Class 4, or Class 4/5.
4. Treatment of LN with twice daily MMF as per the decision of the treating physician.

   The subject will have taken MMF as prescribed by their treating physician for a minimum of 4 days (or 8 doses).
5. Subject tolerates MMF as per the treating physician's opinion;
6. Able to swallow MMF tablets and capsules;
7. If subject is treated with belimumab, must be IV or SQ;
8. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures;
9. Evidence of a personally signed and dated Informed Consent document and Assent document (as appropriate) indicating that the subject and a legally acceptable representative/ parent(s)/legal guardian has been informed of all pertinent aspects of the study.
10. Parent or legal guardian must have a smart phone available and able to support the PLUMM smart phone application.
11. Must be able to complete study questionnaires in English or Spanish.

Exclusion Criteria:

1. Perceived or stated inability to adhere to the study protocol;
2. Hypersensitivity to MMF or any component of the drug product;
3. Presence of features (from SLE or other chronic disease) that a-priori suggest that the subject benefits from other therapies than that suggested or allowable by the study protocol; These disease features include but are not limited to severe, progressive, or uncontrolled hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurologic disease.
4. History of other kidney disease besides LN or prior to the diagnosis of SLE;
5. Need for renal replacement therapy within 2 weeks from Baseline Subjects can have required short-term renal replacement therapy prior to Baseline, for example due to preceding acute kidney injury.
6. Infections:

   1. Untreated latent or active tuberculosis (TB);
   2. Chronic infections requiring treatment;
   3. A subject known to be infected with Human Immunodeficiency Virus (HIV), Hepatitis B;
   4. Diagnosis of any infection requiring hospitalization, parenteral antimicrobial therapy or judged to be opportunistic by the investigator within 4 weeks prior to Baseline visit;
   5. Any treated infections within 2 weeks of Baseline visit;
   6. History of infected joint prosthesis with prosthesis still in situ;
7. Blood dyscrasias, including:

   1. Hemoglobin <8.5 g/dL or Hematocrit <22%;
   2. White Blood Cell count <2.6 x 109/L;
   3. Neutrophil count <1.2 x 109/L;
   4. Platelet count <100 x 109/L;
   5. Lymphocyte count <0.5 x 109/L.
8. 8) Estimated glomerular filtration rate [GFR] <40 mL/min/1.73 m2 calculated using the CKiD U25 equation (see Appendix 4);
9. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the upper limit of normal;
10. Vaccinated or exposed to a live or attenuated vaccine within the 4 weeks prior to Baseline visit;
11. History or current symptoms suggestive of lymphoproliferative disorders (e.g., Epstein Barr Virus [EBV] related lymphoproliferative disorder, lymphoma, leukemia, myeloproliferative disorders, or multiple myeloma);
12. Current malignancy or history of any malignancy with the exception of adequate treated or excised basal cell or squamous cell or cervical cancer in situ;
13. Recent (within 4 weeks prior to Baseline visit) significant trauma or major surgery;
14. Herbal supplements with pharmaceutical properties must be discontinued at least 1week prior to Baseline visit, unless there are sufficient data available regarding the duration of an herbal medication's pharmacokinetic and pharmacodynamic effects to allow a shorter or longer washout to be specified (e.g., 5 half-lives).
15. Oral or intravenous cyclophosphamide must be discontinued 12 weeks prior to Baseline visit
16. Use of prohibited prescription medication as listed in Appendix 3 within the specified time frame prior to Baseline visit
17. Participation in other studies involving investigational drug(s) within 4 weeks or 5 half-lives (whichever is longer) prior to Baseline visit and/or during study participation; Exposure to investigational biologics should be discussed with the Sponsor.
18. Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children and female subjects of childbearing potential who are unwilling or unable to use two highly effective methods of contraception or are abstinent for the duration of the study;
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of MMFPK therapy to the efficacy of MMFBSA therapy | 26 week
  the percentage of subjects achieving at least partial remission of LN (PRR) as per the adapted ACR/EULAR Criteria at Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Hermine I Brunner, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (19):
- United States (19):
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Emory Children's Center, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medicine- Comer Children's, Chicago, Illinois
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Children's Hospital at Montefiore, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine Pediatric Immunology Allergy Rheumatology, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital/University of Washington, Seattle, Washington
  - Children's Wisconsin/Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor fulfills its commitment to publicly disclose clinical trial results through posting the results of studies on ClinicalTrials.gov, or EudraCT, and/or www.cincinnatichildrens.com, and other public registries in accordance with applicable local laws/regulations.
  In all cases, study results are reported by the Sponsor regardless of the outcome of the study. Every effort will be made to report the basic results within 1 year of the end of the trial. Results will be posted at www.clinicaltrials.gov/.
  For all publications relating to the study, the institution and investigators will comply with recognized ethical standards concerning publications and authorship, including Section II - "Ethical Considerations in the Conduct and Reporting of Research" of the Uniform Requirements for Manuscripts Submitted to Biomedical Journals, http://www.icmje.org/index.html#authorship.
  A Publication Committee will be established to oversee publication of the results.
Time Frame: within one year for
Access Criteria: results are available to the public
URL: http://www.clinicaltrials.gov